CLINICAL TRIAL: NCT03494049
Title: Veil-preserving Versus Standard Holmium Laser Enucleation of the Prostate: Randomized Clinical Trial
Brief Title: Veil Preserving HoLEP vs. Stanadard HoLEP
Acronym: MansprostIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP.19.11.49
Record Dates: First submitted 2018-03-31; First posted 2018-04-11 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Post Prostatectomy Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Veil sparring HoLEP (Active Comparator): Early mucosal incision lateral to the Veru followed by early separation of the adenoma from the sphincter ring after identification of the plane of enucleation, this minimizes sphincter stretch.
  Furthermore, more proximal incision of the 12 O'clock mucosal strip sparring a veil of mucosa covering the sphincter ring.
  Interventions: Procedure: Veil sparring HoLEP
- Standard HoLEP (Active Comparator): Standard HoLEP TECHNIQUE as described by Elhilali et al 2010
  Interventions: Procedure: Standard HoLEP

INTERVENTIONS:
Procedure: Veil sparring HoLEP — Early mucosal incision; lateral to the Veru and proximal to the apical bulge of the adenoma, followed by early separation of the adenoma from the sphincter ring after identification of the plane of enucleation, this minimizes sphincter stretch.
  Furthermore, more proximal incision of the 12 O'clock mucosal strip sparring a veil of mucosa covering the sphincter ring.
  Other Names: early apical separation
  Arms: Veil sparring HoLEP
Procedure: Standard HoLEP — Holmium laser enucleation of the prostate in the standard approach described by Elhilali et al 2010
  Arms: Standard HoLEP

SUMMARY:
Postoperative transient stress urine leakage following Holmium laser enucleation of the prostate is one of the problems that frustrate both surgeon and patients

Standard HoLEP might be associated with some stretch of the sphincter and de-epithelization of the sphincter area anteriorly.

In Veil preserving HoLEP, early separation of the adenoma from the sphincter ring minimizes sphincter stretch. Furthermore, more proximal incision of the 12 O'clock mucosal strip sparring a veil of mucosa covering the sphincter ring.

Our hypothesis is that by this technique the early postoperative transient urine leak would be minimized and duration of leakage if anny would be shortened.

DETAILED DESCRIPTION:
Postoperative transient stress urine leakage following Holmium laser enucleation of the prostate is one of the problems that frustrate both surgeon and patients.

Many reports addressed different variables for the cause of post HoLEP urine leakage. Looking for a procedure done by a single surgeon who had tremendous experience of this procedure may enable investigators to identify precisely technical points of interest that may affect post HoLEP stress urine incontinence.

Standard HoLEP might be associated with some stretch of the sphincter and de-epithelization of the sphincter area anteriorly.

In Veil preserving HoLEP, early separation of the adenoma from the sphincter ring minimizes sphincter stretch. Furthermore, more proximal incision of the 12 O'clock mucosal strip sparring a veil of mucosa covering the sphincter ring.

Investigators' hypothesis is that by this technique the early postoperative transient urine leak would be minimized and duration of leakage if any would be shortened.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥50 years
2. ASA (American society of anesthesiologists) score ≤3.
3. TRUS estimated weight ≥40 grams.

Exclusion criteria:

Patients who have any of the following were excluded:

1. Patient with neurological disorder which might affect bladder function as cerebrovascular stroke or Parkinson disease.
2. Active urinary tract infection.
3. Presence of bladder cancer (within the last 2 years).
4. Prostate cancer patients.
5. Patients with bleeding tendency, ongoing anticoagulants or antiplatelet medications
6. Previous prostate surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate surgeries
Enrollment: 180 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
urine incontinence | 1 month postoperative
  one hour pad test for post prostatectomy incontinence, scale from 0 to 4, the higher the more incontinence

SECONDARY OUTCOMES:
international prostate symptom score | 1 year
  Symptoms core assessment, score from 0 to 35, the higher the worse the urinary symptoms
urine flow rate | 1 year
  rate of urine flow per unit time, how many milliliters of urine passed per second, above 15ml/second is normal
urine incontinence | 4 months postoperative
  one hour pad test for post prostatectomy incontinence, scale from 0 to 4, the higher the more incontinence
International Consultation on Incontinence Questionnaire Short-Form | one month postoperative
  Continence core assessment, score from 0 to 21, the higher the worse the urinary continence

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshal, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No